CLINICAL TRIAL: NCT07334015
Title: Assessment of Modified Lip Repositioning Surgery and Z Plasty Frenectomy for Treatment of Excessive Gingival Display
Brief Title: Treatment of Excessive Gingival Display (Lip Repositioning and Z Plasty)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Leen somaf, Dr, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/857
Record Dates: First submitted 2025-12-10; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Excessive Gingival Display

STUDY DESIGN:
Intervention Model Description: 2 groups 16 patient in each group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group: z plasty frenectomy (Experimental): Participants in the study group will be treated with Z- plasty frenectomy and will be followed up for 9 months
  Interventions: Procedure: z plasty frenectomy
- control group : modified lip repositioning (Experimental): Participants in the control group will undergo modified lip repositioning with a follow-up period of 9 months.
  Interventions: Procedure: Modified lip repositioning

INTERVENTIONS:
Procedure: z plasty frenectomy — Z-plasty frenectomy is a surgical procedure in which the frenum is released and rearranged using a Z-shaped incision. This technique helps improve tissue mobility and reduce tension. The procedure is performed under local anesthesia"
  Other Names: Z Plasty
  Arms: study group: z plasty frenectomy
Procedure: Modified lip repositioning — "Modified lip repositioning is a minimally invasive surgical technique used to reduce excessive gingival display. The procedure involves removing a small strip of mucosa and repositioning the upper lip to limit its upward movement during smiling. It is performed under local anesthesia ."
  Other Names: lip repositioning; gummy smile
  Arms: control group : modified lip repositioning

SUMMARY:
evaluate clinically the postoperative outcomes of the Z plasty frenectomy technique in comparison to modified lip repositioning surgery

DETAILED DESCRIPTION:
Excessive gingival display is a cosmetic problem where it is usually managed by different approaches such as lip repositioning.

Aim: Is to evaluate clinically the postoperative outcomes of the Z plasty frenectomy technique in comparison to modified lip repositioning surgery Methodology: The clinical study will include 16 patients with gummy smile divided into two groups equally and randomly according to technique using www.randomizer.org.

Group 1: will be treated with conventional modified lip repositioning technique and the labial frenum will be left intact.

Group 2: will be treated with z plasty frenectomy. Clinical follow up will be at 1,3, 6 and 9 months.

Clinical evaluation will be done through using (VAS). It will be used to measure patient satisfaction through pain killer scale . - Likert scale to measure patient satisfaction - Periodontal probe will be used to measure the relapse. Also signs of infection will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 to 30 years
* ASA physical status I or II
* Presence of excessive gingival display (gummy smile)
* Indication for surgical treatment of excessive gingival display
* Willingness to participate and attend follow-up visits

Exclusion Criteria:

* Poor oral hygiene
* Patients with active acute infection
* Patients with poor oral habits
* Pregnant or lactating women
* Heavy smokers
* Alcohol or drug addicts

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-11-19 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Gingival Display (mm) | Up to 9 months
  Gingival display will be assessed in millimeters using standardized clinical photographs taken at maximum smile. Measurements will be performed using a periodontal probe to determine the vertical distance between the inferior border of the upper lip and the gingival margin of the maxillary central incisors. A reduction in gingival display indicates improvement, while an increase indicates relapse. Measurements will be recorded at baseline and during follow-up visits.

SECONDARY OUTCOMES:
Pain score | Up to 9 months
  Postoperative pain will be assessed using a Visual Analog Scale (VAS) ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Lower scores indicate less pain.
Patient Satisfaction Score | Up to 9 months
  Patient satisfaction will be evaluated using a numerical rating scale from 0 to 10, where 0 indicates complete dissatisfaction and 10 indicates maximum satisfaction. Higher scores indicate greater satisfaction.
Signs of infection | Up to 9 months
  Postoperative infection will be assessed clinically based on the presence of signs such as redness, swelling, pain, discharge, or delayed healing at the surgical site. The outcome will be recorded as present or absent.
Surgical Time | During surgery
  Surgical time will be measured in minutes from the initial incision to the completion of wound closure. Shorter surgical time indicates a more efficient procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

REFERENCES:
- [Background] Tatakis DN. Lip Repositioning Techniques and Modifications. Dent Clin North Am. 2022 Jul;66(3):373-384. doi: 10.1016/j.cden.2022.02.002. Epub 2022 Jun 1. PMID 35738733
- See also: Reference describing the modified lip repositioning surgical technique used to reduce excessive gingival display in gummy smile patients. — https://pubmed.ncbi.nlm.nih.gov/26054167/
- See also: Study explaining the use of Z-plasty for lengthening the upper lip and improving esthetic outcomes in cases of excessive gingival display. — https://pubmed.ncbi.nlm.nih.gov/33655255/